CLINICAL TRIAL: NCT05977608
Title: The Impact of a Telephone Reminiscence Program on Reminiscence Functions and Mental Health Outcomes in Community-Dwelling Older Adults
Brief Title: The Impact of a Telephone Reminiscence Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: StoriiCare Company (Unknown)
Responsible Party: Principal Investigator, Juliette Shellman, Associate Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H23-0046
Record Dates: First submitted 2023-07-12; First posted 2023-08-04 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Mental Health; Loneliness; Social Isolation
MeSH Terms: conditions — Psychological Well-Being; Social Isolation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Participants will be asked to participate in the reminiscence program during the first 6 weeks of the study.
  Interventions: Behavioral: Telephone Reminiscence Intervention
- Group 2 (Experimental): Participants will be asked to participate in the reminiscence program during the second 6 weeks of the study.
  Interventions: Behavioral: Telephone Reminiscence Intervention

INTERVENTIONS:
Behavioral: Telephone Reminiscence Intervention — Participants will receive automatic calls three times a week asking their life experiences and personal memories. They can share as much or as little as they would like. They have up to 10 minutes to record their answer and can end the call at any time by hanging up.They will be able to share the stories online with their families if they want.

SUMMARY:
The purpose of this study is to better understand how a telephone reminiscence program impacts reminiscence functions and mental health outcomes in community-dwelling older adults.This study will take 12 weeks to complete and will include approximately 90 study participants. Participants will be randomly assigned to one of two telephone reminiscence groups.They will be either assigned to begin a telephone reminiscence program immediately or in 6 weeks. Participants will receive automatic calls three times a week asking the meaningful questions about their lives. At week 1, week 6, and week 12, participants will also be asked to complete assessments via phone, by research assistants using four questionnaires.

DETAILED DESCRIPTION:
The prevalence of social isolation and loneliness among older adults is a public health problem. It is reported that 25 % of community-dwelling older adults 65 and older are socially isolated while 43 % of older adults 60 and older feel lonely (Cudge et al., 2020). Research has shown that social isolation and loneliness are associated with cardiovascular disease, stroke, depression, dementia, and mortality (Holjlerda, 2016). Loneliness, in particular, has been identified as a potential predictor of mild cognitive impairment (Bundy, et al., 2021; Sutin et al., 2018; Dahlberg, 2021). As a result of the prevalence data, gerontologists and researchers have cited the need for developing, implementing and testing innovative interventions to address this problem. Reminiscence is one example of a cost-effective intervention shown to decrease loneliness and improve mental health and wellness.

STORII is a telephone reminiscence program designed to provide a service that automatically calls older adults three times a week asking them meaningful questions about their lives. The participants have the opportunity to select curated prompts that enable them to record their life stories through the phone. The participants can choose to share them online with their families. Through formative evaluation of the program, the STORII team has noted that their participants to be highly satisfied and highly engaged. As a result of these informal data, it was decided that a more in-depth investigation should be undertaken. Therefore, the purpose of this study is to examine the impact of the STORII program on reminiscence functions and mental health outcomes in community-dwelling older adults.

Participants will be invited to join a telephone reminiscence program designed to provide a service that automatically calls older adults three times a week asking them meaningful questions about their lives. Examples of the questions are "What is the best meal you have ever tasted?", "What is one of your proudest moments?", "What is your earliest memory?". Participants can share as much or as little as they would like. They have up to 10 minutes to record the answers and can end the call at any time by hanging up. There will be no operator on the line that can hear or respond. The participants can choose to share their stories online with their families.

All outcome measures will be assessed at baseline (T0), 6-week post-test (T1), and at 12-week follow-up (T2). Participants will complete assessments via phone, by trained research assistants using four questionnaires. Assessments will be completed by research assistants who are not aware of participants' allocation.

ELIGIBILITY:
Inclusion Criteria:

* Adults age >60 years;
* English speaking
* Community-dwelling
* Willing to participate in a 12 week study
* Willing and able to share memories using a telephone, 10 minutes, 3 times a week

Exclusion Criteria:

* Significant hearing loss
* Cognitive impairment

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2023-06-25 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Mental health as measured by mean changes in the Mental Health Continuum Short Form (MHC-SF) scores | Baseline, Week 6 (Endpoint), Week 12 (Follow up)
  The Mental Health Continuum Short Form (MHC-SF) (Keyes, 2002) will be used to assess mental health and well-being. The 14 item scale measures emotional, social, and psychological dimensions of mental health. Participants answer each item on a 6-point scale, ranging from 0 and 5, resulting in a total score between 0 to 70. The emotional well-being subscale has a range from 0 to 15, the social well-being subscale scores range from 0 to 25, and the psychological well-being subscale scores range from 0 to 30. Higher scores on MHC- SF indicate a higher level of mental well-being. The MHC-SF has demonstrated excellent internal consistency (>.80) and discriminant validity in adults in the United States (Keyes, 2005, 2006), and its test-retest reliability has also been demonstrated, with an average of 0.68 over three consecutive three-month periods and 0.65 over a 9-month period (Lamers et al., 2011).

SECONDARY OUTCOMES:
Change in reminiscence functions as measured by mean changes in the Modified Reminiscence Functions Scale (MRFS) scores | Baseline, Week 6 (Endpoint), Week 12 (Follow up)
  The Modified Reminiscence Functions Scale (MRFS) containing 29 items will be used to measure reminiscence functions. The scale measures the frequency of different reminiscence functions identified as: (a) self-regard, (b) death preparation, (c) bitterness revival, (d) conversation, and (e) intimacy maintenance, teach and inform, boredom reduction, and conversation. Respondents are asked to report their level of agreement with statements such as, "When I reminisce, it is to teach younger people about cultural values" or "When I reminisce, recalling my past help me know who I am now" on a 5-point scale ranging from 1 (never) to 5 (very often). A higher score indicates more frequent reminiscences for the specific function. The Cronbach's Alpha for the subscales ranged from .73 to .91, indicating good internal consistency (Shellman & Zhang, 2014; Washington, 2009).
Change from loneliness as measured by mean changes in UCLA 3 Item Loneliness Scale scores | Baseline, Week 6 (Endpoint), Week 12 (Follow up)
  UCLA 3 Item Loneliness Scale (UCLA 3) (Russell, 1996) is a brief 3-item scale that measures three dimensions of loneliness: relational connectedness, social connectedness, and self. Responses are provided on a 3-point response scale ranging from "hardly" to "often", with total scores ranging from 3 to 9. Higher scores indicate a higher level of loneliness. The instrument has favorable psychometric properties, including high internal consistency (ranging from 0.89 to 0.94) and a good test-retest reliability over one year (r = .73) (Russell, 1996).
Change from life satisfaction as measured by mean changes in the Satisfaction with Life Scale scores | Baseline, Week 6 (Endpoint), Week 12 (Follow up)
  The Satisfaction with Life Scale (SWLS) (Diener et al., 1985) is a measure of life satisfaction that includes five statements, such as "In most ways, my life is close to my ideal." Responses are provided on a seven-point scale ranging from (1) "strongly disagree" to (7) "strongly agree", with a total score ranging from 7 to 35. Higher scores indicate greater life satisfaction. The scale is a highly reliable measure, with good internal consistency (0.87) and high test-retest reliability over a 2-month period (r = .82) (Diener et al., 1985).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keyes CL. The mental health continuum: from languishing to flourishing in life. J Health Soc Behav. 2002 Jun;43(2):207-22. PMID 12096700
- [Background] Diener E, Emmons RA, Larsen RJ, Griffin S. The Satisfaction With Life Scale. J Pers Assess. 1985 Feb;49(1):71-5. doi: 10.1207/s15327752jpa4901_13. PMID 16367493
- [Background] Russell DW. UCLA Loneliness Scale (Version 3): reliability, validity, and factor structure. J Pers Assess. 1996 Feb;66(1):20-40. doi: 10.1207/s15327752jpa6601_2. PMID 8576833
- [Background] Shellman JM, Zhang D. Psychometric testing of the Modified Reminiscence Functions Scale. J Nurs Meas. 2014;22(3):500-10. doi: 10.1891/1061-3749.22.3.500. PMID 25608435
- [Background] Cudjoe TKM, Roth DL, Szanton SL, Wolff JL, Boyd CM, Thorpe RJ. The Epidemiology of Social Isolation: National Health and Aging Trends Study. J Gerontol B Psychol Sci Soc Sci. 2020 Jan 1;75(1):107-113. doi: 10.1093/geronb/gby037. PMID 29590462